CLINICAL TRIAL: NCT03600870
Title: A Phase 1 Proof-of-concept Clinical Trial Evaluating the Safety and Tolerability of Midodrine in Hepatopulmonary Syndrome
Brief Title: Midodrine in Hepatopulmonary Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hilary M. DuBrock,, Assistant Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-006221
Record Dates: First submitted 2018-06-20; First posted 2018-07-26 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hepatopulmonary Syndrome (HPS)
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): All subjects enrolled will be assigned to receive midodrine. The initial starting dose will be midodrine 5mg orally three times a day. After 7-10 days, patients will increase the dose to 10mg three times a day as tolerated if no adverse effects occur. Treatment duration will be 6 months.
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Midodrine is an oral alpha-1 agonist that increases vascular tone. It is administered orally. The initial starting dose will be midodrine 5mg orally three times a day. After 7-10 days, patients will increase the dose to 10mg three times a day as tolerated if no adverse effects occur. Treatment duration will be 6 months.

SUMMARY:
This proof-of-concept clinical trial will determine the safety and tolerability of midodrine in patients with hepatopulmonary syndrome (HPS). Exploratory endpoints will assess the effect of midodrine on oxygenation, intrapulmonary shunting and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to very severe hepatopulmonary syndrome, defined as the presence of all of the following:

  1. Liver disease or portal hypertension
  2. Intrapulmonary shunting on contrast-enhanced echocardiogram
  3. Hypoxemia [A-a gradient ≥15mmHg (or ≥20mmHg if age >64) and PaO2<80mmHg on arterial blood gas testing]
* Ability to provide informed consent
* Ability to comply with study medication use and testing, in the opinion of the principal investigator or co-investigator

Exclusion Criteria:

* Vulnerable study population, including imprisoned individuals, non-English speaking patients
* Participation in other investigational drug studies
* Any of the following conditions:
* Systolic blood pressure>160mmHg or diastolic blood pressure >100mmHg
* Heart rate <50bpm
* Urinary retention at baseline
* Left ventricular ejection fraction <50%
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Women of child-bearing potential not willing or able to use highly effective methods of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events (AEs)) | 6 months
  Outcome will be defined by the incidence of adverse events (AEs) that occur during the study period. An adverse event is defined as any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Abnormal results of diagnostic procedures are considered to be AEs if the abnormality results in study withdrawal, is associated with a serious AE, is associated with clinical signs or symptoms, leads to additional treatment or further diagnostic tests or is considered by the investigator to be of clinical significance. Each adverse event will be further characterized by severity and relationship to the study drug. Adverse event are classified as serious if they are: fatal, life-threatening, require or prolongs hospital stay, lead to persistent or significant disability or incapacity or a congenital anomaly or birth defect.

SECONDARY OUTCOMES:
Arterial Oxygenation | 3 months and 6 months
  Describe the effect of midodrine on:
  • arterial oxygenation (PaO2 and A-a gradient )(mmHg)
Diffusion capacity | 3 months and 6 months
  Describe the effect of midodrine on:
  • percent predicted diffusion capacity for carbon monoxide (Range 0-100%)
Cardiac output | 3 months and 6 months
  Describe the effect of midodrine on cardiac output (L/min) as estimated by echocardiogram in patients with HPS.
Intrapulmonary shunting | 3 months and 6 months
  Describe the effect of midodrine on severity (mild, moderate or severe) of intrapulmonary shunting (as assessed by echocardiogram shunt study) in patients with HPS.
Intrapulmonary shunting | 6 months
  Describe the effect of midodrine on severity of intrapulmonary shunting (as assessed by percent shunt index (0-100%) on technetium macroaggregated albumin scan) in patients with HPS.
Symptoms as assessed by Modified Medical Research Council (MMRC)dyspnea scale | 3 months and 6 months
  Describe the effect of midodrine on MMRC dyspnea scale (0-4). Higher numbers indicate more severe dyspnea.
6 minute walk distance | 3 months and 6 months
  Describe the effect of midodrine on 6 minute walk distance, in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary M DuBrock, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials